CLINICAL TRIAL: NCT00527839
Title: Prospective Evaluation of the Clinical and Economic Outcomes of Total Joint Replacement: HSS Shoulder Arthroplasty Cohort
Brief Title: Hospital for Special Surgery Shoulder Arthroplasty Cohort
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-014
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Total joint replacements are some of the most successful medical devices developed over the last fifty years. They enable millions of people to remain ambulatory and pain free, with minimal risk. In 2002, over 200,000 total hip replacements, 350,000 total knee replacements, and 25,000 total or partial shoulder replacements were performed in the United States (HCUP data). Future use will likely be even higher: it is estimated that by the year 2020, the population 65 and over in developed countries will increase by 71%. Existing studies do not provide adequate prospective data to evaluate long-term outcomes.

HSS is a world leader in total joint replacement including total shoulder arthroplasty. However, there is no systematic follow-up or evaluation of patients who have their shoulders replaced here.

The purpose of this study is to establish a prospective cohort of HSS total shoulder arthroplasty to evaluate predictors of outcome, causes of failure and to allow ongoing evaluation of the results of our patients over time.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and undergoing total shoulder arthroplasty at HSS

Exclusion Criteria:

* No other exclusion criteria. Pregnant women are eligible for the registry as this is a non-interventional study which only involves filling out questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will be asking all patients undergoing a total shoulder arthroplasty to participate.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-04; Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome Measures (PROMs) | Collection of at Baseline, 6 Months, 1 Year, 2 Year, 5 Year and 10 Year
  Patient reported outcomes (PROMs) at 1 year, 2 year, 5 year, 10 year follow-up time points. This information will be collected and maintained for use in future research studies with their own individually defined outcomes.
Intra Operative Data | Collection of data on Day 0 (Date of Surgery)
  Surgeon reported data
Demographic data | Collection of at Baseline, 6 Months, 1 Year, 2 Year, 5 Year and 10 Year
  Collection of patient information and demographic data

CONTACTS AND LOCATIONS:
Overall Officials: Robert Marx, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- See also: CERTS tools and resources — http://www.certs.hhs.gov